CLINICAL TRIAL: NCT05284409
Title: Comparative Study Between the Prophylactic Intravenous Administrations of Acetaminophen vs Dexamethasone vs Pethidine Regarding the Incidence of Shivering Induced by Single Shot Spinal Anesthesia in the Orthopedic Surgeries of the Lower Limbs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Nouh, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ADP
Record Dates: First submitted 2022-02-28; First posted 2022-03-17 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Shivering
MeSH Terms: interventions — Meperidine; Acetaminophen; Dexamethasone

STUDY DESIGN:
Intervention Model Description: The assigned medication will be prepared in a color coded 250 ml polypropylene bottle of normal saline. The administration of the assigned infusion will be done by a resident not involved in the study after stabilization of the sensory blockade level over a duration of 15 to 20 minutes, the study drugs will be prepared by the hospital pharmacy and follow-up of the patients will be conducted by the anesthesia residents not involved in any other part of the study.
  Group A: (control group) 36 patients will receive 0.5 mg/kg Pethidine IVI for management of shivering induced by Single Shot Spinal Anesthesia.
  Group B: 36 patients will receive 15 mg/kg Acetaminophen IVI for management of shivering induced by Single Shot Spinal Anesthesia.
  Group C: 36 patients will receive 0.1 mg/kg Dexamethasone IVI for management of shivering induced by Single Shot Spinal Anesthesia.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pethidine (Active Comparator): (control group) 36 patients will receive 0.5 mg/kg Pethidine IVI for management of shivering induced by Single Shot Spinal Anesthesia.
  Interventions: Drug: Pethidine
- Acetaminophen (Experimental): 36 patients will receive 15 mg/kg Acetaminophen IVI for management of shivering induced by Single Shot Spinal Anesthesia.
  Interventions: Drug: Acetaminophen
- Dexamethasone (Experimental): 36 patients will receive 0.1 mg/kg Dexamethasone IVI for management of shivering induced by Single Shot Spinal Anesthesia.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Pethidine — 36 patients will receive 0.5 mg/kg Pethidine IVI
  Arms: Pethidine
Drug: Acetaminophen — 36 patients will receive 15 mg/kg Acetaminophen IVI
  Arms: Acetaminophen
Drug: Dexamethasone — 36 patients will receive 0.1 mg/kg Dexamethasone IVI
  Arms: Dexamethasone

SUMMARY:
Single Shot Spinal anesthesia (SSSA) is associated with considerable perioperative shivering and can be challenging to treat. Some pharmacologic agents like N-methyl d-aspartate receptor antagonists, magnesium sulfate and opioid analgesics have been used for restriction of post-spinal anesthesia shivering. Besides that shivering is poorly understood, the gold standard for the treatment and prevention has not been defined yet.

This study is to determine the effect of prophylactic intravenous administration of acetaminophen versus dexamethasone versus pethidine in controlling shivering induced by spinal anesthesia

DETAILED DESCRIPTION:
Aim of this study is to compare between the prophylactic intravenous administrations of acetaminophen vs dexamethasone vs pethidine regarding the incidence of shivering induced by single shot spinal anesthesia in the orthopedic surgeries of the lower limbs

Ethical Considerations: Approval of the research ethical committee of the faculty of medicine, Ain Shams University will be obtained and informed written consents will be taken from all the participants after full clarification of the study and their rights for withdrawal at any time will be assured and their privacy will be guaranteed. The single shot spinal anesthesia technique will be performed by a single experienced anesthetist.

Study tools: Bedside Shivering Assessment Scale (BSAS) to indicate the degree of shivering at the time of its onset either intra or postoperatively, and throughout the duration of one hour at the post-anesthesia care unit (PACU).

Study Interventions: The study will include 108 patients fulfilling the inclusion criteria undergoing orthopedic surgeries of the lower limbs. The patients will be randomized into three equal groups by a computer-generated table of random numbers, each including 36 patients, namely groups A, B, and C according to the drug used as an anti-shivering agent. The assigned medication will be prepared in a color coded 250 ml polypropylene bottle of normal saline. The administration of the assigned infusion will be done by a resident not involved in the study after stabilization of the sensory blockade level over a duration of 15 to 20 minutes, the study drugs will be prepared by the hospital pharmacy and follow-up of the patients will be conducted by the anesthesia residents not involved in any other part of the study.

Group A: (control group) 36 patients will receive 0.5 mg/kg Pethidine IVI for management of shivering induced by Single Shot Spinal Anesthesia.

Group B: 36 patients will receive 15 mg/kg Acetaminophen IVI for management of shivering induced by Single Shot Spinal Anesthesia.

Group C: 36 patients will receive 0.1 mg/kg Dexamethasone IVI for management of shivering induced by Single Shot Spinal Anesthesia.

All patients will be assessed preoperatively, and will be instructed to fast for 6 hours.

On arrival to the operating theatre, all patients will have an inserted peripheral wide bore IV access (18 G). Anti-stress measures: intravenous pantoprazole 40 mg will be given. I.V. fluids will be preheated to room temperature. Lactated Ringer's solution will be infused at 10 ml/kg over 30 min before spinal anesthesia. The infusion rate will then be modified according to the intraoperative fluid balance.

Conventional monitoring including electrocardiogram (ECG), heart rate (HR), non-invasive blood pressure (NIBP) and pulse oximetry (SPO2) will be conducted. Hemodynamic readings (Mean arterial blood pressure (MAP), HR, and SPO2), peripheral and room temperatures will be recorded before the administration of the single shot spinal anesthesia. The operating and recovery rooms temperatures will be maintained at 25°C±1 with approximately 60% humidity.

Preoperatively, all of the patients will receive titration of 0.5 mg Midazolam increments on intravenously as an anesthetic adjuvant. Anesthetic equipment and drugs for resuscitation will be kept ready at hand before starting the spinal anesthesia. Supplemental oxygen (6 liter/min) will be administered via a facemask during the operation.

The patients in all of the groups will receive SSSA. The blocks will be performed by well trained personnel. The blocks will be performed before administration of the compared medications after obtaining intravenous (IV) access and application of standard ASA monitoring. Under complete aseptic conditions, single shot spinal anesthesia will be instituted at either L3/4 or L4/5 interspaces. 2.8 mL (14 mg) of 0.5% hyperbaric bupivacaine at a rate of 0.2 ml/sec will be injected in the sitting position by an anesthetist who was blind to the study by using 25 gauge Quincke spinal needle. The patient will be placed in the Supine position. The sensory blockade level will be checked in order not to reach the level of T4.

Sensory levels will be assessed by pinprick test to determine the peak sensory level and time to two segment regression in minutes. Motor block will be assessed by using Modified Bromage scale (16) (0 = no block 1 = hip block, 2 = hip and knee block, 3 = hip, knee, and ankle block) to determine the time to reach complete motor block and duration of motor blockade (in minutes).

The desired motor and sensory block will be Bromage scale 3 and T6, respectively.

All of the patients will be covered with one layer of surgical drapes over the chest, thighs, and calves during the operation and one cotton blanket over the entire body after operation. Assessment parameters: HR, MAP, and SPO2 will be recorded using standard non-invasive monitors before intrathecal injection and thereafter at 5, 10, 15, 20 minutes then every 10 minutes to complete 90 minutes from the intrathecal injection.

All of the patients will be observed for: Hypotension (defined as a decrease in MAP of more than 20% from baseline or a decrease of the systolic arterial blood pressure below 90 mmHg and baseline MAP will be calculated from three measurements taken in the ward before the operation) will be treated by crystalloid infusion and if necessary ephedrine 5 mg IV will be administered. The amount of ephedrine given in each group will be recorded. Bradycardia will be considered if the heart rate is less than 50 beats/min and will be treated with IV atropine (0.01mg/kg).

Pruritus will be assessed by a four-point ordinal scale where zero points to no itching, one points to mild itching, two points to moderate itching, treatment not requested, three points to severe itching, treatment requested.

In case of pruritus (45.5 mg intramuscular pheniramine hydrogen maleate) will be given.

The administration of the assigned infusion will be done by a resident not involved in the study after stabilization of the sensory blockade level over the duration of 15 to 20 minutes.

The level of sedation will be assessed according to a five-point range: [1] alert and oriented, [2] somnolent, [3] closed eyes, arousable on a verbal order, [4] closed eyes, arousable to physical stimuli and [5] closed eyes and patient unarousable to physical stimuli.

Body temperature (axillary temperature) will be recorded with a percutaneous thermometer. The ambient temperature will be measured by a wall thermometer. The ambient temperature will be maintained at 25 degree Celsius with constant humidity. Fluid management intraoperatively will be done according to bodyweight of the patient and intra-operative losses.

When shivering occurs, it will be graded using Bedside Shivering Assessment Scale (BSAS): 0 - None: No Shivering, 1 - Mild: Shivering localized to neck/thorax, maybe seen only as artifact on ECG or felt by palpation 2 - Moderate: Intermittent involvement of the upper extremities +/- thorax 3 -Severe: Generalized shivering or sustained upper / lower extremity shivering.

In all of the groups, the degree of shivering will be assessed at the time of its onset either intra or postoperatively, and throughout the duration of one hour at the post-anesthesia care unit (PACU). Grade 3 or 4 of shivering score will be regarded as failure of prophylaxis, and a rescue dose of 0.2 mg/kg Pethidine IV will be administered and the total dose will be recorded.

Patients will be admitted to the PACU. Patient's satisfaction will be assessed by asking the patient to answer the question, "How would you rate your experience after the operation?" using a 7-point Likert verbal rating scale, and acceptable satisfaction score of the patient will range from 5 to 7 (1 - Extremely dissatisfied, 2 - Dissatisfied, 3 - Somewhat dissatisfied, 4 - Undecided, 5 - Somewhat satisfied, 6 - Satisfied, 7 - Extremely satisfied).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA) I or II.
* Both sexes.
* Age ranging from 20 to 55 years old.
* Body weight ranging from 60 to 100 kilograms.
* Receiving Single Shot Spinal anesthesia.
* Scheduled for orthopedic surgeries of the lower limb.

Exclusion Criteria:

* Patient's refusal.
* Allergy to local anesthetics or any of the studied drugs.
* Patients with significant cognitive dysfunction.
* Duration of surgery more than 120 min.
* Patients with hypo- or hyperthyroidism.
* An initial body temperature >38.0 or <36.0 degree Celsius.
* Receiving vasodilators, or medications likely to alter thermoregulation.
* Pregnancy.
* Sensory blockade level reaching T4 or higher.
* Obesity (BMI > 35 kg/m2).

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The incidence of shivering | During procedure to up to one hour at the post-anesthesia care unit (PACU)
  The incidence of shivering induced by single shot spinal anesthesia after the prophylactic administration of the study medications.
  When shivering occurs, it will be graded using Bedside Shivering Assessment Scale (BSAS): 0 - None: No Shivering, 1 - Mild: Shivering localized to neck/thorax, maybe seen only as artifact on ECG or felt by palpation 2 - Moderate: Intermittent involvement of the upper extremities +/- thorax 3 -Severe: Generalized shivering or sustained upper / lower extremity shivering.
  In all of the groups, the degree of shivering will be assessed at the time of its onset either intra or postoperatively, and throughout the duration of one hour at the post-anesthesia care unit (PACU). Grade 3 or 4 of shivering score will be regarded as failure of prophylaxis, and a rescue dose of 0.2 mg/kg Pethidine IV will be administered and the total dose will be recorded.

SECONDARY OUTCOMES:
The need to administer pethidine | The time of administration of pethidine
  In all of the groups, the degree of shivering will be assessed at the time of its onset either intra or postoperatively, and throughout the duration of one hour at the post-anesthesia care unit (PACU). Grade 3 or 4 of shivering score will be regarded as failure of prophylaxis, and a rescue dose of 0.2 mg/kg Pethidine IV will be administered.
the total dose of Pethidine given | The time of administration of pethidine
  In all of the groups, the degree of shivering will be assessed at the time of its onset either intra or postoperatively, and throughout the duration of one hour at the post-anesthesia care unit (PACU). Grade 3 or 4 of shivering score will be regarded as failure of prophylaxis, and a rescue dose of 0.2 mg/kg Pethidine IV will be administered and the total dose will be recorded.
The patient's satisfaction | up to one hour postoperative
  Patient's satisfaction will be assessed by asking the patient to answer the question, "How would you rate your experience after the operation?" using a 7-point Likert verbal rating scale, and acceptable satisfaction score of the patient will range from 5 to 7 (1 - Extremely dissatisfied, 2 - Dissatisfied, 3 - Somewhat dissatisfied, 4 - Undecided, 5 - Somewhat satisfied, 6 - Satisfied, 7 - Extremely satisfied).
The level of sedation | within 5 minutes after the administration of sedative
  The level of sedation will be assessed according to a five-point range: [1] alert and oriented, [2] somnolent, [3] closed eyes, arousable on a verbal order, [4] closed eyes, arousable to physical stimuli and [5] closed eyes and patient unarousable to physical stimuli.
Pruritus | during procedure
  Severity of pruritus. Pruritus will be assessed by a four-point ordinal scale where zero points to no itching, one points to mild itching, two points to moderate itching, treatment not requested, three points to severe itching, treatment requested.

CONTACTS AND LOCATIONS:
Overall Officials: Galal A Al Kadi, MD, Study Director — Professor of Anesthesia
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No